CLINICAL TRIAL: NCT00074971
Title: A Multi-center, Open-Label Extension Study of the Safety and Efficacy of Recombinant Human a-Galactosidase A (r-haGAL) Replacement in Patients With Fabry Disease
Brief Title: A Study of the Safety and Efficacy of Fabrazyme in Patients With Fabry Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Coporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGAL-005-99
Record Dates: First submitted 2003-12-24; First posted 2003-12-25 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Fabry Disease
Keywords: a-Galactosidase A; aGAL; r-haGAL; Fabry; GL-3; Fabrazyme
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase beta

INTERVENTIONS:
Drug: Fabrazyme (agalsidase beta)

SUMMARY:
People with Fabry disease have an alteration in their genetic material (DNA) which causes a deficiency of the a-galactosidase A enzyme. Fabrazyme is a drug that helps to breakdown and remove certain types of fatty substances called "glycolipids." These glycolipids are normally present within the body in most cells. In Fabry disease, glycolipids build up in various tissues such as the liver, kidney, skin, and blood vessels because a-galactosidase A is not present, or is present in small quantities. The build up of glycolipid ("globatriaosylceramide" or "GL-3") levels in these tissues in particular is thought to cause the clinical symptoms that are common to Fabry disease. This study will test the safety and efficacy of Fabrazyme in the treatment of patients with Fabry disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have successfully completed the previous double-blind study (AGAL-1-002-98)
* Patients must provide written informed consent prior to study participation
* Female patients must have a negative pregnancy test prior to each dosing and use a medically accepted method of contraception throughout the study

Exclusion criteria:

* Patient has undergone kidney transplant or is currently on dialysis
* Patient is pregnant or lactating
* Patient is unwilling to comply with the requirements of the protocol
* Patient has a clinically significant organic disease (with the exception of symptoms related to Fabry disease), including clinically significant cardiovascular, hepatic, pulmonary, neurologic, or renal disease, or other medical condition, serious intercurrent illness, or extenuating circumstances that, in the opinion of the investigator, would preclude participation in the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58
Dates: Start 1999-10; Study Completion 2004-12

PRIMARY OUTCOMES:
Safety and efficacy
Morphologic assessment of GL-3 inclusions in the capillary endothelium (vasculature) of the kidney

SECONDARY OUTCOMES:
Changes in McGill Pain Questionnaire
Autonomic status
Glomerular filtration
Functional assessment of urinary protein excretion Ophthalmic changes
SF-36 Health Survey
Physician's assessment of Fabry Symptoms and pain medication

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme Coorporation
Locations (20):
- United States (14):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California San Fransisco, San Francisco, California
  - Northwest Oncology & Hematology Associates, Coral Springs, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Fetal Diagnostic and Imaging Center, Billings, Montana
  - University of New Mexico, Albuquerque, New Mexico
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester School of Medicine, Rochester, New York
  - Hart Family Practice, Hickory, North Carolina
  - Hematology/Oncology Associates of South Texas, San Antonio, Texas
  - University of Washington School of Medicine, Seattle, Washington
- France (2):
  - Hospital Edouard Herriot, Lyon
  - Hospital Europeen Georges Pompidou, Paris
- Academisch Medisch Centrum, Amsterdam, Netherlands
- University of Puerto Rico, San Juan, Puerto Rico
- United Kingdom (2):
  - National Hospital for Neurology and Neurosurgery, London
  - Hope Hospital, Manchester

REFERENCES:
- [Derived] Germain DP, Charrow J, Desnick RJ, Guffon N, Kempf J, Lachmann RH, Lemay R, Linthorst GE, Packman S, Scott CR, Waldek S, Warnock DG, Weinreb NJ, Wilcox WR. Ten-year outcome of enzyme replacement therapy with agalsidase beta in patients with Fabry disease. J Med Genet. 2015 May;52(5):353-8. doi: 10.1136/jmedgenet-2014-102797. Epub 2015 Mar 20. PMID 25795794